CLINICAL TRIAL: NCT05494632
Title: Effects of Interaural Frequency and Loudness Mismatch on SSD-CI Performance
Brief Title: Interaural Frequency and Loudness Mismatch in SSD CI Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Cochlear (Industry)
Responsible Party: Principal Investigator, Jill B Firszt, PhD, Professor, Washington University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202206085
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-06

CONDITIONS: Outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Period 1: Study 1 (Experimental): CI speech processor programming in experienced cochlear implant (CI) recipients with single sided deafness. Program changes were made to decrease the interaural frequency mismatch between the CI ear and the contralateral ear.
  Interventions: Device: Treatment-modifications to CI speech processor program. Specifically reducing interaural frequency mismatch in experienced SSD-CI recipients.
- Period 2: Study 2 (Experimental): CI speech processor programming in newly implanted cochlear implant (CI) recipients with single sided deafness. Program changes were made to decrease the interaural frequency mismatch between the CI ear and the contralateral ear.
  Interventions: Device: Treatment-modifications to CI speech processor program to reduced interaural frequency mismatch in newly implanted SSD-CI recipients.
- Period 3: study 3 (Experimental): CI speech processor programming in experienced cochlear implant (CI) recipients with single sided deafness. Program changes were made to decrease the interaural loudness mismatch between the CI ear and the contralateral ear.
  Interventions: Device: Treatment-modifications to CI speech processor program to reduced interaural loudness mismatch in experienced SSD-CI recipients.

INTERVENTIONS:
Device: Treatment-modifications to CI speech processor program. Specifically reducing interaural frequency mismatch in experienced SSD-CI recipients. — We will modify the CI speech processor program to reduce interaural frequency mismatch between the CI ear and the contralateral ear in experienced CI recipients with SSD.
  Arms: Period 1: Study 1
Device: Treatment-modifications to CI speech processor program to reduced interaural frequency mismatch in newly implanted SSD-CI recipients. — We will modify the CI speech processor program to reduce interaural frequency mismatch between the CI ear and the contralateral ear in newly implanted CI recipients with SSD.
  Arms: Period 2: Study 2
Device: Treatment-modifications to CI speech processor program to reduced interaural loudness mismatch in experienced SSD-CI recipients. — We will modify the CI speech processor program to reduce interaural loudness mismatch between the CI ear and the contralateral ear in experienced CI recipients with SSD.
  Arms: Period 3: study 3

SUMMARY:
Interaural loudness and pitch mismatch in single-sided deaf cochlear implant (SSD-CI) recipients reduces binaural processing cues and contributes to performance outcomes, specifically speech understanding in noise and localization. The study aims to improve binaural cues through speech processor program modifications that reduce interaural mismatches.

DETAILED DESCRIPTION:
Effective binaural processing depends on similar loudness growth functions at each ear. The use of interaural level differences (ILDs), perceived as loudness differences, to locate sound is critical given the inability of cochlear implant (CI) recipients to use interaural time differences (ITDs) in binaural processing. In CI recipients with single-sided deafness (SSD), perceived interaural loudness differences may not be valid indicators of interaural level differences because the CI compresses amplitude. Studies suggest better preservation of ILDs may contribute to improved localization and understanding in noise. Since SSD-CI recipients use only one device, an approach to improve their use of ILDs is to match perceived loudness at each ear.

Binaural processing is also affected when signals of equal frequency are not matched in pitch at each ear. In bilateral CI recipients, the investigators found that the greater the pitch mismatch between ears, the poorer the speech understanding in noise. The investigators want to extend this work to SSD-CI recipients. Through CI program modifications, the study aims to decrease the pitch and loudness mismatch between the CI ear and the normal hearing ear to improve binaural listening abilities, specifically speech understanding in noise and sound localization.

ELIGIBILITY:
Inclusion Criteria:

* Participants for the proposed study will be adults with single-sided deafness. Participants will have at least 6 months experience with their cochlear implant or will be newly implanted with the cochlear implant.

Inclusion criteria for the experienced CI user group and the newly implant group are as follows:

* 18 years of age and older
* Postlingual onset of SSD
* Pure tone average (PTA) at 500, 1000, and 2000 Hz of less than or equal to 30 dB HL in the contralateral ear, known as the normal hearing ear
* Implanted with or chosen to be implanted with a Nucleus cochlear implant
* Full insertion of electrode array

Exclusion Criteria:

* • Not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill B Firszt, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from July of 2022 through 2023.
Pre-assignment Details: In Study 2, 5 participants used the default FAT for 6 weeks, then used the modified FAT for 6 weeks. 5 other participants used the modified FAT for 6 weeks, then the default FAT for 6 weeks. This was done to prevent order effects. Finally, all participants compared both FATs for 2 weeks. All 10 participants were tested twice with each FAT.
Groups:
- Period 1: Study 1: For twenty experienced single-sided deaf (SSD) cochlear implant (CI) participants, we compared their everyday frequency allocation table (FAT) in their speech processor program to a modified FAT. The modified FAT attempted to reduce interaural frequency mismatch between the CI ear and the contralateral ear.
- Period 2: Study 2 Group Starting With Default FAT: For 5 newly implanted SSD-CI participants, the manufacturer's default frequency allocation table (FAT) was compared to a modified FAT that attempted to reduce interaural frequency mismatch between the CI ear and the contralateral ear. Five participants were assigned the default FAT at initial activation of the device.
- Period 2: Study 2 Group Starting With Modified FAT: For 5 newly implanted SSD-CI participants, a modified frequency allocation table (FAT) was compared to the manufacturer's default FAT. The modified FAT attempted to reduce interaural frequency mismatch between the CI ear and the contralateral ear. Five participants were assigned the modified FAT at initial activation of the device.
- Period 3: Study 3: For fifteen participants, we compared their everyday speech processor program with a modified loudness program. The modified program was created to reduce the interaural loudness mismatch between the CI ear and the normal hearing ear in these experienced CI recipients with SSD.
Period: Overall Study
Arm/Group | Period 1: Study 1 | Period 2: Study 2 Group Starting With Default FAT | Period 2: Study 2 Group Starting With Modified FAT | Period 3: Study 3
Started | 20 | 5 | 5 | 15
Completed | 20 | 5 | 5 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants in study 1 & 2 were experienced SSD-CI users. Participants in study 2 were new SSD-CI recipients with no CI experience. Per study protocol, half began CI use with the default FAT and half with the modified FAT, switching FATs after 6 wks use & finally comparing both FATs on the CI processor. Data of interest are results between the 2 FATs. Results of participants who used the default FAT 1st and those who used the modified FAT 1st are not of interest and therefore weren't analyzed.
Groups:
- Period 1: Study 1: For 20 participants, we compared their everyday frequency allocation table (FAT) in their CI speech processor program to a modified FAT. The modified FAT was created to reduce the interaural frequency mismatch between the CI ear and the contralateral ear of experienced CI recipients with single sided deafness (SSD). Participants were tested twice with each FAT over about an 8-10 week period. Speech recognition in noise was the primary result analyzed.
- Period 2: Study 2 Group Starting With Default FAT: For 5 newly implanted participants, we compared the manufacturer's default frequency allocation table (FAT) in their CI speech processor program to a modified FAT. The modified FAT was created to reduce the interaural frequency mismatch between the CI ear and the contralateral ear of newly implanted CI recipients with single sided deafness (SSD). Five participants were assigned the default FAT at initial activation of the device. Participants were tested twice with each FAT over about a 16 week period. Speech recognition in noise was the primary result.
- Period 2: Study 2 Group Starting With Modified FAT: For 5 newly implanted participants, we compared a modified FAT to the manufacturer's default FAT in their CI speech processor program. The modified FAT was created to reduce the interaural frequency mismatch between the CI ear and the contralateral ear of newly implanted CI recipients with single sided deafness (SSD). Five participants were assigned the modified FAT at initial activation of the device. Participants were tested twice with each FAT over about a 16 week period. Speech recognition in noise was the primary result.
- Period 3: Study 3: For 15 participants, we compared their everyday speech processor program to a modified speech processor program. The modified program was created to reduce the interaural loudness mismatch between the CI ear and the normal hearing ear in these experienced CI recipients with SSD. Participants were tested twice with each program, i.e., their everyday program and the modified loudness program over about an 8-10 week period. Speech recognition in noise was the primary result.
- Total: Total of all reporting groups
Arm/Group | Period 1: Study 1 | Period 2: Study 2 Group Starting With Default FAT | Period 2: Study 2 Group Starting With Modified FAT | Period 3: Study 3 | Total
Number analyzed (Participants) | 20 | 5 | 5 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 4 | 5 | 7 | 29
  >=65 years | 7 | 1 | 0 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (10.8) | 49.6 (13.0) | 56.8 (12.6) | 61.7 (10.9) | 58.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 4 | 11 | 28
  Male | 9 | 3 | 1 | 4 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 20 | 3 | 5 | 14 | 42
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Speech Understanding in Noise, Measured With the R-Space Test Environment. The R-Space Test Environment Simulates Speech Understanding in a Noisy Restaurant.
Description: Participants speech understanding was evaluated in the R-Space test environment with two speech processor programs, an everyday or default program and a modified program. The modified program was created to reduce interaural frequency or loudness mismatch between participants' CI ear and normal hearing ear. The R-Space simulates listening in a noisy restaurant, a real-world listening situation. The score is a signal-to-noise ratio that reflects 50% speech understanding in noise. Participants are surrounded by 8 loudspeakers with restaurant noise from all 8. A sentence is presented from the front loudspeaker. Participants repeat back what they hear. The noise is adjusted adaptively. For a correct response, the noise is increased; it is decreased for an incorrect response. This provides signal-to-noise ratio (SNR) for 50% speech understanding. The average score for participants with normal hearing is -5 dB SNR. A lower number represents better performance than a higher number.
Time Frame: Participants were tested in the R-Space twice with each speech processor program, e.g., everyday or default program and modified program. The testing was carried out within a 2-3 month time period, and after using each program for at least 6 weeks.
Population: 20 experienced SSD-CI participants were tested in the R-Space with their everyday use FAT and with the modified FAT (Study 1). Ten newly implanted SSD-CI participated in Study 2. The newly implanted group were tested in the R-Space with the manufacturer's default FAT and with a modified FAT. Fifteen experienced SSD-CI users were tested in the R-SPACE with their everyday program and with a modified loudness program (Study 3). Testing was done twice with each FAT or loudness program.
Measure: Median (Standard Deviation); unit: signal-noise-ratio in decibels (dB)
Groups:
- Period 1: Study 1: Twenty experienced single-sided deaf cochlear implant recipients (SSD-CI) compared their everyday speech processor program frequency allocation table (FAT) to a modified FAT. The modified FAT was created to reduce interaural frequency mismatch between the normal hearing ear and the cochlear implant ear. Participants were first tested with their everyday FAT. They were tested a second time after 6 weeks use of the modified FAT. Lastly, they compared both FATs on their speech processor at home for several weeks, after which they were tested a second time with each FAT.
- Period 2: Study 2 Group starting with default FAT: Five newly implanted single-sided deaf cochlear implant recipients (SSD-CI) participated. They compared the manufacturer's default FAT to a modified FAT. The modified FAT was created to reduce interaural frequency mismatch between the normal hearing ear and the cochlear implant ear. Five participants were assigned the manufacturer's default FAT at initial activation. After 6 weeks use of the default FAT, participants were tested and then began using the modified FAT for another 6 weeks. Participants were tested with the modified FAT at the end of six weeks. Then, participants compared FATs on their speech processor for several weeks and were tested with each FAT a second time.
- Period 2: Study 2 Group starting with Modified FAT: Five newly implanted single-sided deaf cochlear implant recipients (SSD-CI) participated. They compared a modified FAT to the manufacturer's default FAT. The modified FAT was created to reduce interaural frequency mismatch between the normal hearing ear and the cochlear implant ear. Five participants were assigned the modified FAT at initial activation. After 6 weeks use of the modified FAT, participants were tested and then began using the default FAT for another 6 weeks. Participants were tested with the default FAT at the end of six weeks. Then, participants compared FATs on their speech processor for several weeks and were tested with each FAT a second time.
- Period 3: Study 3: Fifteen experienced SSD-CI recipients compared their everyday speech processor program to a modified loudness speech processor program. The modified loudness program was created in an attempt to balance loudness between the normal hearing ear and the cochlear implant ear and therefore decrease interaural loudness mismatch. Participants were first tested with their everyday program. They were tested a second time after 6 weeks use of the modified program. Lastly, they compared both programs on their speech processor at home for several weeks, after which they were tested a second time with each program.
Arm/Group | Period 1: Study 1 | Period 2: Study 2 Group starting with default FAT | Period 2: Study 2 Group starting with Modified FAT | Period 3: Study 3
Number analyzed (Participants) | 20 | 5 | 5 | 15
signal-noise-ratio in decibels (dB)
  Everyday FAT (study 1), Default FAT (study 2), Everyday loudness program (study 3) | -3.0 (1.6) | -1.9 (1.9) | -4.0 (0.7) | -2.9 (1.1)
  Modified FAT (study 1 and 2), Modified loudness program (study 3) | -3.6 (1.1) | -2.9 (2.5) | -3.6 (1.0) | -4.1 (1.0)
Statistical Analysis 1: Comparison: Period 1: Study 1; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — the threshold for statistical significance was <=0.05; Median Difference (Net) = 1.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of approximately 16 weeks for each group.
Description: Adverse events were not formally collected during this study. However, all-cause mortality and serious adverse were monitored due to the fact that the participants came to a number of test sessions and the researchers would have been aware if a serious adverse event would have occurred. No serious adverse events took place during this study.
Groups:
- Period 2: Study 2: Ten newly implanted single-sided deaf cochlear implant recipients (SSD-CI) participated. They compared the manufacturer's default FAT to a modified FAT. The modified FAT was created to reduce interaural frequency mismatch between the normal hearing ear and the cochlear implant ear. Five participants were assigned the manufacturer's default FAT at initial activation. Five were assigned to the modified FAT at initial activation. After 6 weeks use of the default or modified FAT, participants were tested and then began using the FAT that they had not been using, for another 6 weeks. Participants were tested again at the end of six weeks. They were tested a third time after comparing both FATs for several weeks.
Arm/Group | Period 1: Study 1 | Period 2: Study 2 | Period 3: Study 3
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10 | 0/15
Other Adverse Events (participants affected / at risk) | 0/20 | 0/10 | 0/15

LIMITATIONS AND CAVEATS:
One of the limitations was the small number of SSD participants in the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT05494632/Prot_SAP_000.pdf